CLINICAL TRIAL: NCT00002791
Title: A PHASE II STUDY OF NEOADJUVANT CHEMOTHERAPY AND RADIATION THERAPY IN THE MANAGEMENT OF HIGH-RISK, HIGH-GRADE, SOFT TISSUE SARCOMAS OF THE EXTREMITIES AND BODY WALL
Brief Title: Chemotherapy Plus Radiation Therapy Followed by Surgery in Treating Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: RTOG-9514; CDR0000064856; E-R9514; RTOG-R9514
Record Dates: First submitted 1999-11-01; First posted 2004-09-02 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Sarcoma
Keywords: stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Filgrastim; Dacarbazine; Doxorubicin; Ifosfamide; Mesna; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: ifosfamide
Drug: mesna
Procedure: conventional surgery
Radiation: brachytherapy
Radiation: intraoperative radiation therapy
Radiation: radioisotope therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy followed by surgery in treating patients who have soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess whether patients with high-grade soft tissue sarcoma (STS) treated with neoadjuvant mesna/doxorubicin/ifosfamide/dacarbazine (MAID) plus radiotherapy in a cooperative group setting exhibit a response rate, toxicity, and complication rate comparable to those seen in pilot data collected by the Massachusetts General Hospital. II. Assess local control and local complications related to surgery and neoadjuvant MAID plus radiotherapy in these patients. III. Develop a tissue repository of frozen STS for ancillary genetic and flow cytometric analysis of these tumors. IV. Form an Intergroup Working Sarcoma Group that will develop a patient base, relationships, and support for the future development and completion of a phase III study of adjuvant therapy for STS.

OUTLINE: The following acronyms are used: DOX Doxorubicin, NSC-123127 DTIC Dacarbazine, NSC-45388 EBRT External-Beam Radiotherapy (equipment unspecified) G-CSF Filgrastim; Granulocyte Colony-Stimulating Factor (Amgen), NSC-614629 IFF Ifosfamide, NSC-109724 MAID Mesna/DOX/IFF/DTIC Mesna Mercaptoethane sulfonate, NSC-113891 3-Drug Combination Chemotherapy plus Radiotherapy followed by Surgery followed, if indicated, by Radiotherapy followed by 3-Drug Combination Chemotherapy. MAID; plus EBRT to the primary tumor and suspected microscopic disease; followed by minimal wide surgical excision; followed, if positive margins, by postoperative EBRT; followed by MAID.

PROJECTED ACCRUAL: There will be 60 patients accrued into this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed soft tissue sarcoma of an extremity or the body wall that is a primary or a postoperatively recurrent tumor Biopsy required within 2 months prior to entry Grade II or III tumor, including AJCC stages IIB and IIIB lesions at least 8 cm in diameter No more than 4 chest lesions that are no greater than 3 mm in diameter on preoperative CT The following histologies are excluded: Angiosarcoma of the scalp or face Chondrosarcoma Extraosseous Ewing's sarcoma Head and neck sarcoma Kaposi's sarcoma Osteosarcoma Primitive neuroectodermal tumor Rhabdomyosarcoma Patients on this study are also eligible for Frozen Tumor Repository study (protocol RTOG-9308)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 80%-100% Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 50 U Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No congestive heart failure (CHF) within 6 months No myocardial infarction (MI) within 6 months No New York Heart Association class II-IV heart disease Left ventricular ejection fraction at least 50% by MUGA or echocardiogram If history of CHF or MI, criterion must be met within past 6 months Other: No contraindication to surgery No uncontrolled bacterial, viral, or fungal infection No serious medical or psychiatric illness that precludes informed consent or limits survival to less than 2 years No second malignancy within 5 years except: Surgically treated in situ cervical cancer Nonmelanomatous skin cancer Not pregnant or nursing Negative pregnancy test required of fertile women within 7 days prior to entry Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-02; Primary Completion 2002-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Kraybill, MD, FACS, Study Chair — Roswell Park Cancer Institute; Ronald H. Blum, MD, Study Chair — NYU Langone Health
Locations (237):
- United States (220):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Urology Associates - Mobile AL, Mobile, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscallosa, Alabama
  - Providence Cancer Therapy Center, Anchorage, Alaska
  - Arizona Cancer Center, Tucson, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mount Diablo Medical Center, Concord, California
  - Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Cancer Care Center, Pomona, California
  - Mercy Medical Center - Redding, Redding, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Santa Cruz Radiation Oncology Medical Group, Inc., Santa Cruz, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford University, Stanford, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Radiation Oncology Center - Walnut Creek, Walnut Creek, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Whittingham Cancer Center, Norwalk, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lykes Center for Radiation Therapy, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - West Florida Cancer Institute - Pensacola, Pensacola, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - InterCommunity Cancer Center at Rome, Rome, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Clarion Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - St. Joseph's Radiation Oncology Center, South Bend, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Medical Center at Bowling Green, Bowling Green, Kentucky
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Western Baptist Hospital, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Romagosa Radiation Oncology Center, Lafayette, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Radiation Oncology Affiliates of Maryland, P.A., Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Joint Center for Radiation Therapy, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Ozarks Regional, Springfield, Missouri
  - Veterans Affairs Medical Center - Saint Louis, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Elizabeth General Medical Center - West, Elizabeth, New Jersey
  - South Jersey Hospital - Millville, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua-Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Saint Joseph Medical Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - Genesee Hospital - Rochester, Rochester, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - UNI-MED Medical Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. John Medical Center, Tulsa, Oklahoma
  - Samaritan Regional Cancer Center, Corvallis, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Penn State Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Catholic Medical Center, Mercy Fitzgerald Divison, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Allegheny University Hospitals- Hahnemann, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Julie and Ben Rogers Cancer Institute, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Green Mountain Oncology Group, Rutland, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Baptist Hospital, Lynchburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Swedish Hospital Tumor Institute, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Oncology Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
- Canada (16):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Kraybill WG, Harris J, Spiro IJ, Ettinger DS, DeLaney TF, Blum RH, Lucas DR, Harmon DC, Letson GD, Eisenberg B. Long-term results of a phase 2 study of neoadjuvant chemotherapy and radiotherapy in the management of high-risk, high-grade, soft tissue sarcomas of the extremities and body wall: Radiation Therapy Oncology Group Trial 9514. Cancer. 2010 Oct 1;116(19):4613-21. doi: 10.1002/cncr.25350. PMID 20572040
- [Result] Kraybill WG, Harris J, Spiro IJ, Ettinger DS, DeLaney TF, Blum RH, Lucas DR, Harmon DC, Letson GD, Eisenberg B; Radiation Therapy Oncology Group Trial 9514. Phase II study of neoadjuvant chemotherapy and radiation therapy in the management of high-risk, high-grade, soft tissue sarcomas of the extremities and body wall: Radiation Therapy Oncology Group Trial 9514. J Clin Oncol. 2006 Feb 1;24(4):619-25. doi: 10.1200/JCO.2005.02.5577. PMID 16446334
- [Result] Kraybill WG, Spiro I, Harris J, et al.: Radiation Therapy Oncology Group (RTOG) 95-14: a phase II study of neoadjuvant chemotherapy (CT) and radiation therapy (RT) in high risk (HR), high grade, soft tissue sarcomas (STS) of the extremities and body wall: a preliminary report. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1387, 2001.
- [Derived] Wang D, Harris J, Kraybill WG, Eisenberg B, Kirsch DG, Ettinger DS, Kane JM 3rd, Barry PN, Naghavi A, Freeman CR, Chen YL, Hitchcock YJ, Bedi M, Salerno KE, Severin D, Godette KD, Larrier NA, Curran WJ Jr, Torres-Saavedra PA, Lucas DR. Pathologic Complete Response and Clinical Outcomes in Patients With Localized Soft Tissue Sarcoma Treated With Neoadjuvant Chemoradiotherapy or Radiotherapy: The NRG/RTOG 9514 and 0630 Nonrandomized Clinical Trials. JAMA Oncol. 2023 May 1;9(5):646-655. doi: 10.1001/jamaoncol.2023.0042. PMID 36995690
- [Derived] Kane JM 3rd, Magliocco A, Zhang Q, Wang D, Klimowicz A, Harris J, Simko J, DeLaney T, Kraybill W, Kirsch DG. Correlation of High-Risk Soft Tissue Sarcoma Biomarker Expression Patterns with Outcome following Neoadjuvant Chemoradiation. Sarcoma. 2018 Feb 28;2018:8310950. doi: 10.1155/2018/8310950. eCollection 2018. PMID 29681762